CLINICAL TRIAL: NCT00484978
Title: A Single Center Prospective Phase II Study: Stereotactic Radiosurgery to the Resection Cavity Following Surgical Removal of Brain Metastasis
Brief Title: Stereotactic Radiosurgery to the Resection Cavity Following Surgical Removal of Brain Metastasis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-056 TASMC
Record Dates: First submitted 2007-06-11; First posted 2007-06-12 (Estimated); Last update posted 2007-06-12 (Estimated); Status verified 2007-06

CONDITIONS: Brain Neoplasms
Keywords: Stereotactic Radiosurgery; Surgery; Metastatic tumor to brain; radiation; Brain Metastases of all pathologies
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stereotactic Radiosurgery

SUMMARY:
Brain metastases (BM) are the most common intracranial tumors in adults and source of the most common neurological complications of systemic cancer. Surgery and radiation therapy are the most important components in the management of BM with the goal to prolong survival and improve the quality of life. Whole brain radiotherapy (WBRT) has shown to increase local and distant control both with and without surgical resection. However, patients who develop a new or recurrent BM after WBRT and undergo resection are left without adjuvant therapy options. Local recurrence particular in patients with single metastasis does effect both survival and quality of life. In individual cases the option of additional radiotherapy has been suggested and applied. We seek to evaluate the addition of a stereotactic radiosurgery (SRS) boost to the resection cavity both as adjuvant and salvage procedure among patients, who undergo resection of a BM and previously received WBRT or decline WBRT. Goal is to show superior local brain control.

DETAILED DESCRIPTION:
Study Purpose

Treatment strategies for recurrent brain metastasis

Limited clinical data support interventions for recurrent BM such as WBRT, re-operation or SRS, depending on previous treatments (6, 45, 48). Two retrospective analyses looked at a total of 130 non-small cell lung cancer (NSCLC) patients with recurrent BM after resection (6, 45). ,Recurrence happened at the original site in approximately two/thirds of the patients and at other sites for the remainders; Re-resection had a significant effect on prolonged survival compared to patients who did not undergo it (p=0.001). A small subgroup of these patients underwent a third resection with a median survival of 42 months. A more recent study looked at resection of BM that had previously been treated with SRS (48). Sixty-one patients with 1-3 previously treated BM recurred and underwent resection. Major neurological morbidity occurred in 2% and no mortality was observed. A multivariate analysis showed that higher RPA class, focal treatment (surgery or SRS), and treatment of new additional lesions significantly affected survival. Re-operation of a previously focally treated BM provided long-term control and positive impact on survival. Additionally, confirming the pathological diagnosis in a recurrent lesion after SRS is important, as radiation necrosis can occur in 2.3%-8.6% of the patients, a condition that requires a different treatment approach than that for recurrent metastasis (5, 10, 14).

Surgery and radiation therapy are important components in the complex treatment of BM and can prolong survival and improve the quality of life. Patients, who develop brain metastasis after WBRT remain with limited options. A resection will diminish the local disease significantly; however adjuvant radiation might further increase the control rate. We plan to evaluate the addition of a stereotactic radiosurgery (SRS) boost to the resection cavity both as adjuvant and salvage procedure in patient, who underwent resection of a BM and previously received WBRT or decline WBRT.

Study Design

The study is designed to observe patients for feasibility, efficacy and toxicity:

Patient Enrollment Informed Consent will be obtained and then eligibility screening will be assessed using Inclusion/ Exclusion criteria. A patient who appears to meet ALL eligibility requirements will be asked to participate in the study.

Variables Measured The primary end point will be evaluated following obtaining follow up neuro-imaging (contrast Brain CT or MRI).

The secondary end points will be measured as follows:

* Evaluation of CT and MRI by neuro-radiologist. - Individual response: comparison between pre-treatment and follow-up MRI performed at 2-3 months intervals or according to clinical indication.
* Side effects during and following the treatment, as well as self reported (or otherwise obtained) absence of side effects.

Pre-Procedure

Screening process:

Patients with known systemic malignancy, who underwent surgical resection of a brain metastasis and fulfill the eligibility criteria specified for this study (see inclusion/exclusion criteria)

Imaging:

All patients will undergo a contrast CT and MRI brain imaging in preparation of the treatment.

Neurological Baseline Assessment:

A standard neurological baseline examination shall take place. The neurological examination will include the following:

* Cognitive function ( Mini Mental Status)
* Cranial nerves
* Motor Strength
* Deep tendon reflexes
* Plantar response
* Sensory
* Coordination/Gait

ELIGIBILITY:
Inclusion Criteria:

* Patient must have undergone surgical resection of a brain metastasis
* Patients with no more than 3 brain metastases on contrast MRI.
* Previous WBRT for brain malignancy, except patients with melanoma, renal cell carcinoma.
* Adult patient aged > 18.
* Patient must be in adequate general health, as indicated by:

  * Karnofsky performance status equal or greater than 60.
  * The absence of a concomitant life-threatening disease other than the malignancy.
* Patient must understand the investigational nature of this study and sign informed consent form, approved by the Institutional Review Board.

Exclusion Criteria:

* Pregnancy
* Patients unable or unwilling to follow protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2007-02; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Improved local tumor control after resection | 6months and 12 months

SECONDARY OUTCOMES:
Overall survival Quality of life | QoL 3-6-12months and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Kanner, MD, Principal Investigator — Tel Aviv Medical Center, affiliated Tel Aviv University
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel